CLINICAL TRIAL: NCT01261195
Title: Establishment of Vascular Permeability Model for Research Purpose by Human
Brief Title: Establishment of Vascular Permeability Model for Research Purpose by Human Umbilical Vascular Endothelial Cells
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Jih-Jin Tsai, Kaohsiung Medical University Chung-Ho Memorial Hospital
Other Study IDs: KMUH-IRB-990030
Record Dates: First submitted 2010-12-14; First posted 2010-12-16 (Estimated); Last update posted 2011-08-17 (Estimated); Status verified 2011-06

CONDITIONS: Healthy People

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — the umbilical cord
Oversight: Data Monitoring Committee: Yes

SUMMARY:
HUVEC primary cells for researches about the relation between plasma leakage and infections.

DETAILED DESCRIPTION:
This study is going to collect HUVEC primary cells to set up an in vitro model for researches about the relation between plasma leakage and infections.

ELIGIBILITY:
Inclusion Criteria:

* healthy pregnant women
* would like to join this study

Exclusion Criteria:

* venereal disease

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: healthy pregnant women
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2010-03; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Jih-Jin Tsai, Doctor, Principal Investigator — KMUH Tropical Medicine Center
Locations (1):
- Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City, Kaohsiung, Taiwan